CLINICAL TRIAL: NCT06844734
Title: Intrathecal Baclofen for the Management of Hereditary Spastic Paraparesis: a Prospective Cohort Study
Brief Title: A Prospective Cohort Study of ITB Treatment for HSP
Acronym: ITB-HSP
Status: Recruiting | Type: Observational
Sponsor: Shanghai 6th People's Hospital (Other)
Responsible Party: Principal Investigator, Li Cao, Professor, Shanghai 6th People's Hospital
Other Study IDs: 2024-KY-305(K)
Record Dates: First submitted 2025-02-10; First posted 2025-02-25 (Actual); Last update posted 2025-02-26 (Actual); Status verified 2025-01

CONDITIONS: Hereditary Spastic Paraplegia
Keywords: Hereditary Spastic Paraparesis; Intrathecal baclofen
MeSH Terms: conditions — Spastic Paraplegia, Hereditary

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Intrathecal baclofen management of hereditary spastic paraparesis: Patients with hereditary spastic paraparesis aged 14 to 70 years, with a Modified Ashworth Scale score of greater or equal to 3 in 2 or more joints of lower limb, and agree to undergo Intrathecal baclofen surgery will be recruited. Patients will receive professional assessment every six months.
- The oral baclofen group: Patients who do not agree to intrathecal baclofen treatment or those who do not achieve satisfactory therapeutic effect during the baclofen testing phase will be included in oral baclofen group. Patients will receive professional assessment every six months, with natural history observation.

SUMMARY:
The investigators conduct a prospective cohort study to explore the treatment effectiveness of continuous infusion of intrathecal baclofen (ITB) for hereditary spastic paraplegia (HSP) in China, delve into the optimal timing for starting treatment, and investigate the response differences among different subtypes. The ultimate goal is to provide clinical evidence and guidance for the application of ITB in treating HSP in China, as well as improve the life expectancy and quality of life for HSP patients. The main questions it aims to answer are:

1. Changes in gait and motor function, as well as spasticity levels, compared to pre-surgery and control group after ITB surgery.
2. Changes in quality of life, pain, psychological and emotional status, and cognition compared to pre-surgery and control group after ITB surgery.
3. Complications following ITB surgery.
4. Impact of ITB surgery on the occurrence and progression of skeletal deformities.
5. Subgroup analysis: comparing surgical outcomes between different genotypes and between simple versus complex types.
6. Determine the optimal timing for ITB intervention.

DETAILED DESCRIPTION:
Hereditary spastic paraplegias (HSPs) are a heterogeneous group of neurodegenerative disorders characterized by progressive spasticity and weakness of the lower limbs due to retrograde axonal degeneration of the corticospinal tract. Baclofen is a selective GABA-B receptor agonist and is commonly used for the treatment of spasticity. Baclofen can be administered orally or intrathecally by the surgical implantation of a specialized pump. Intrathecal baclofen (ITB) is significantly more potent for the treatment of spasticity than the oral form. The goal of this clinical trial is to explore the efficacy and safety of ITB in the treatment of HSP patients. This study is prospective, open-label, single center, and this trial will last for 3 years. A total of 50 patients will participate. Twenty-five patients who will receive ITB and the other 25 control patients will receive oral baclofen. Patients with HSP aged 14 to 70 years, with a Modified Ashworth Scale score of ≥3 in ≥2 joints of lower limb, will be recruited. Patients who do not agree to undergo ITB and/or those who have an inadequate response during intrathecal baclofen test will receive oral baclofen therapy and undergo natural history observation. Professional clinical evaluations are conducted regularly for both groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients meet the clinical and genetic diagnostic criteria of hereditary spastic paraplegia (HSP);
* Age: 14 to 70 years old
* Modified Ashworth Score for lower limbs: ≥2 joints with muscle tone ≥grade 3
* Patients are willing to participate in clinical trials and able to understand and comply with the research program

Exclusion Criteria:

* Patients are allergic to the baclofen
* Other neurological diseases likely affecting the evaluation of study treatment
* Other medical conditions such as: heart disease, tumor, blood disease, liver disease, kidney disease, etc. in the past 1 year
* Pregnancy or lactating women or subjects who are unable to use appropriate contraception during the trial
* Participating in another study drug trial and used the investigational drug in the past 30 days
* Subjects have poor compliance or other factors that are not suitable for participating in the clinical trial

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients meet the clinical and genetic diagnostic criteria of hereditary spastic paraplegia (HSP) between 14 to 70 years old with of lower limbs. Participants suffered from severe spasticity with score ≥ 3 by Modified Ashworth assessment in ≥2 joints of lower limbs. Patients agree to participate in clinical trials and able to understand and comply with the research program.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-03-01 (Estimated)

PRIMARY OUTCOMES:
Six-Minute Walk Test(6-MWT) | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  The 6-MWT measures the distance a person can walk in six minutes. A shorter distance indicates lower exercise capacity.
Step length | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Step length is measured by gait analysis device. Step length refers to the distance from the heel strike of one foot to the heel strike of the opposite foot. Longer step length indicates that the patient has improved lower limb muscle strength and coordination, and that spastic symptoms have been alleviated.
walking speed | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Walking speed is measured by gait analysis device. Walking speed refers to the distance covered by a person within a unit of time while walking, expressed in meters per minute (m/min). An increase in walking speed indicates an improvement in spasticity and motor function.
knee flexion angle | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Knee flexion angle is measured by gait analysis device.An increase in the knee flexion angle indicates improved motor function and reduced spasticity.
Modified Ashworth Scale(MAS) | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  range: 0-4, higher scores mean more severe spasticity.
Range of Motion (ROM) of Joints | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  ROM refers to the distance and direction a joint can move to its full potential. Flexion, extension, abduction, adduction of joints are measured.

SECONDARY OUTCOMES:
Patient Global Impression of Change (PGIC) scale | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  range (1-7), lower scores mean a better outcome
Oswestry Disability Index (ODI) | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  The ODI consists of 10 sections (items). Each section is scored on a scale of 0 to 5, with higher scores indicating greater levels of disability.
Numeric Rating Scale (NRS) | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  rang 0 to 10, higher scores mean a worse outcome
MMSE score | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Mini-Mental State Examination (MMSE) : range: 0-30, higher scores mean a better outcome
MoCA score | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Montreal Cognitive Assessment (MoCA) score: range: 0-30, higher scores mean a better outcome.
SDS | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Self-Rating Depression Scale: Index score < 50 Normal range; 50-59 Mild depression; 60-69 Moderate depression; ≥70 Severe depression
SAS | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Self-Rating Anxiety Scale (SAS): 20-44 Normal range; 45-59 Mild to moderate anxiety levels; 60-74 Marked to severe anxiety levels; 75 and above Extreme anxiety levels
SPRS score | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  The change in the Spastic Paraplegia Rating Scale (SPRS) score : range: 0-52, higher scores mean a worse outcome
Complications | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Catheter breakage, blockage, infection, etc.
GMFM-88 | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Gross Motor Function Measure-88 (GMFM-88) score: range: 0-264, higher scores mean a better outcome
GAS | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Goal Attainment Scale (GAS) - Family Goal Selection Version: range: -2-+2, higher scores mean a better outcome
Foot deformity molding | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Utilizing CT digital 3D reconstruction technology
Scoliosis assessment | From the end of treatment to observations at 6 months, 12months, 18months, 24months, 30months, and 36months respectively
  Measurement of the Cobb angle using spinal X-ray imaging

CONTACTS AND LOCATIONS:
Overall Officials: Li Cao, phD, Principal Investigator — Shanghai Jiao Tong University Affiliated Sixth People's Hospital
Locations (1):
- Shanghai Sixth People's Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No